CLINICAL TRIAL: NCT01240018
Title: Probiotics and Satiety - Acute Effects and Persistence of Acute Effects
Brief Title: ProSat - Long Term Effect of Probiotics on Satiety
Acronym: ProSat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B257II
Record Dates: First submitted 2010-06-25; First posted 2010-11-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Appetite Regulation
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotic
- High dose Lb. casei (Active Comparator)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Parallel, randomized, controlled 2 arms study.

SUMMARY:
The aim of the ProSat study is to examine the effects of a probiotic capsule containing Lb. Casei on subjective appetite sensation, ad libitum energy intake, and appetite hormone response in a single meal test and to determine whether the acute effects persist after daily supplementation of the probiotic capsule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Normal to slight overweight (BMI: 22-28 kg/m2)
* 20-45 years of age

Exclusion Criteria:

* Smoking
* Daily medicine use (oral contraceptives excluded)
* Use of pre- and probiotic supplements and foods
* Blood donation 3 months prior to the study
* Hb < 7,5mmol/l
* Chronic illnesses such as hyperlipidemia, diabetes inflammatory diseases
* Pregnancy or breastfeeding
* Elite athletes (>10 hours hard exercise/week)
* Vegetarians

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Glucose, insulin, GLP-1, GLP-2, CCK, PYY, PP, ghrelin, amylin, LPS, TNF-alfa, CRP, fibrinogen. | June 2011

SECONDARY OUTCOMES:
Subjective appetite measurements, spontaneous food intake. | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MD, Principal Investigator — Department of Human Nutrition, Copenhagen University, Denmark
Locations (1):
- University of Copenhagen, Department of Human Nutrition, Frederiksberg, DK, Denmark